CLINICAL TRIAL: NCT05481450
Title: A Prospective, Randomized, Double-Blind, Parallel, Placebo-Controlled, Clinical Interventional Study to Evaluate the Efficacy and Safety of Nutritears® in Adult Subjects With Dry Eye Syndrome
Brief Title: Efficacy and Safety Safety of Nutritears® in Adults With Dry Eye Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: True Eye Experts - New Tampa (Unknown); True Eye Experts - Lutz (Unknown); True Eye Experts - South Tampa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OA051022
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blind, parallel, placebo-controlled, clinical interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Experimental): Consume one capsule every morning after the breakfast at the same time every day for 56 days
  Interventions: Dietary Supplement: Nutritears®
- Placebo (Placebo Comparator): Consume one capsule every morning after the breakfast at the same time every day for 56 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritears® — Strength: Lutein/Zeaxanthin - 20/4 mg; Curcuminoids 200 mg; Vitamin D3 600 IU (Total capsule weight ≈670 mg)
  Arms: Dietary supplement
Dietary Supplement: Placebo — Soybean oil capsule (Total capsule weight ≈670 mg)
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, parallel, placebo-controlled, clinical interventional study. The purpose of this study is to evaluate the efficacy and safety of Nutritears®, a dietary supplement of OmniActive Health Technologies, in adult subjects with dry eye syndrome (DES). Subjects shall be instructed to consume one capsule of their assigned investigational study product every morning after the breakfast, at the same time every day, for 56 days (8 weeks).

DETAILED DESCRIPTION:
Dry eye syndrome (DES) affects a significant population around the world. Tear film moistens and prevents the ocular surface from dust, toxins, pollutants, etc. An imbalance in any of the tear film layers accompanied by glandular dysfunction leads to DES and it affects the ocular surface. The symptoms include discomfort, visual disturbance, inflammation, damage to ocular surface and tear film instability. This is a prospective, randomized, double-blind, parallel, placebo-controlled, clinical interventional study. The purpose of this study is to evaluate the efficacy and safety of Nutritears®, a dietary supplement of OmniActive Health Technologies, in adult subjects with dry eye syndrome (DES).

After the informed consent process, completion of all screening assessments and once all the inclusion/exclusion criteria are met, the eligible subjects shall be enrolled in the study. Medical history, including a complete review of all current and past diseases and their respective treatments, will be performed during the screening visit. Physical examination including detailed ocular examination and vital signs (like blood pressure, pulse rate, oxygen saturation and body temperature) will be done during screening. Interviews will be conducted to assess/obtain the medical history, ophthalmic history, systemic disease history, current occupation, exposure to air, presence of allergic problems or concomitant systemic diseases, topical and systemic medications, spectacles/contact lens usage, oral contraceptives, significant history of trauma, chemical burns, drug reactions, history of using any kind of tear substitute, other connective tissue disorder and any history of ocular surgery shall be obtained. Digital screen exposure time from devices like computers, laptops, televisions, tablets, and mobile phones will be recorded.

The following screening tests and procedures shall also be conducted on each potential subject prior to consideration for inclusion into the study:

If the clinical signs and symptoms of DES are present, the following test shall be performed on both the eyes of each subject.

1. Schirmer's Test
2. Ocular Surface Disease Index (OSDI)
3. Tear Film Break-Up Time (TBUT)
4. Standard Patient Evaluation of Eye Dryness (SPEED)
5. Corneal and Conjunctival Staining
6. Tear Osmolarity
7. MMP-9 biomarker

If the subject is eligible as per the inclusion/exclusion criteria then, at Randomization Visit, subjects will be randomly (Double-blind) assigned in 1:1 ratio to one of the two (2) treatment groups i.e., Nutritears® or Placebo at Visit 2.

Subjects will be instructed to consume one capsule every morning after the breakfast, at the same time every day, for 56 consecutive days (8 weeks).

Subjects shall complete five scheduled clinic visits as follows:

* Visit 1: Screening Visit (Day -7 to Day -1) • Visit 2: Randomization Visit (Day 1)
* Visit 3: First Follow-Up Visit (Day 14 ± 3 days)
* Visit 4: Second Follow-Up Visit (Day 28 ± 3 days)
* Visit 5: End of Treatment Visit (Day 56 + 3 days) Total study duration for the clinical part shall be a maximum of 66 days which includes the screening period of 7 days, followed by the treatment period of 56 (8 weeks) and an End of study visit at 56 + 3 days.

Safety assessments include monitoring of adverse events (AEs), physical examination, vital signs (heart rate, blood pressure, oxygen saturation, body temperature) and laboratory assessments. Clinical assessments include the Schirmer's Test, Ocular Surface Disease Index (OSDI), Tear Film Break-Up Time (TBUT), Standard Patient Evaluation of Eye Dryness (SPEED) and Corneal and Conjunctival Staining, Tear Osmolarity and MMP-9 biomarker.

A subject diary shall be provided to the subjects to record the Investigational Product administration details, rescue medication (artificial tears) usage, side effects, and concomitant medication details. All subjects shall be instructed to complete the subject diary after each investigational study product administration. Any additional and missed administrations should also be noted in the subject diary. The daily dosing data shall be used to evaluate compliance. Statistical comparisons for therapeutic efficacy shall be made between Nutritears® to the Placebo product.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects aged between 18 and 65 years (both limits inclusive).
2. Clinical diagnosis of symptomatic Dry Eye Syndrome confirmed by a licensed optometrist at Baseline by presence of irritation, foreign body (sandy) sensation, feeling of dryness, itching, non-specific ocular discomfort and altered/effected QoL at least in any one of the eyes.
3. Subjects shall be in good health and free from any clinically significant disease, other than Dry Eye Syndrome (DES), that might interfere with the study evaluations.
4. Subjects must meet the following criteria in at least one eye, as determined by a licensed optometrist:

   i. Schirmer's Test without anesthesia ≤ 10 mm ii. Ocular Surface Disease Index (OSDI) Test symptoms between 12 and 40
5. Subjects with any of the following in at least one eye, as determined by a licensed optometrist:

   i. Tear film break up time ≤ 10 seconds ii. Tear Osmolarity ≥ 316 milliosmole /L iii. Fluorescein corneal staining ≥ 1 and < 3.
6. Subject willing to provide written consent.
7. Subjects shall be willing and able to understand and comply with the requirements of the study, administer the study product as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study.

Exclusion Criteria:

1. Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
2. History of allergy or sensitivity to Lutein, Zeaxanthin, Curcumin or Vitamin D3, related compounds or any component of the formulation.
3. Presence of severe dry eye syndrome with complications such as perforated Corneal Ulcer, Uveitis and Glaucoma, in the Investigator's opinion that may interfere with the evaluation of the Subject's Dry Eye Syndrome (DES).
4. Current evidence of ocular infections or inflammatory conditions like acute conjunctivitis or other medical condition that, in the Investigator's opinion, would place the Subject at undue risk by participating or compromise the integrity of the study data.
5. Subject with poorly controlled diabetes mellitus, rheumatoid arthritis and Systemic Lupus Erythematosus (SLE) which causes Dry Eye Syndrome.
6. Subjects with herpetic eye disease.
7. Subjects with chronic infection of the lacrimal gland.
8. Subjects with Laser In Situ Keratomileusis (LASIK).
9. Subjects with poorly controlled hypertension (>140/96 mm of Hg).
10. Subjects with evidence of malignancy.
11. Subjects suffering from major systemic illness necessitating long term drug treatment (Psychological, Neurological, Endocrinal, Cardiovascular disorders, etc.).
12. Subjects with concurrent serious Hepatic Dysfunction or Renal Dysfunction, uncontrolled Pulmonary Dysfunction (asthmatic and Chronic Obstructive Pulmonary Disease (COPD) Subjects) or other concurrent severe disease.
13. Any ocular trauma or surgery that may affect corneal sensitivity and/or normal tear distribution (e.g., cataract surgery, refractive surgery) within the 6 previous months to study inclusion
14. Subjects with inability to swallow soft gel capsules.
15. Use of lutein, zeaxanthin, curcumin, or vitamin D3 on prescription for other medical indications or for health-conscious reasons
16. Use of steroids or hormone replacement therapy or any other medication that may adversely affect the outcome of the study.
17. Subjects on aspirin or anti-coagulant therapy.
18. Subjects with any other medical condition that might adversely impact the safety of the study participants or confound the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Schirmer's Test (without anesthesia) | Baseline, Day 14, Day 28, Day 56
  Change from Baseline in the length of wetting on a sterile Schirmer's Test strip.
  Without previously instilling anesthetic drops, the Schirmer strip is inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding touching the cornea, and the length of wetting strips in millimeters is recorded after 5 minutes. The patients will be instructed to close their eyes gently. After 5 minutes have elapsed, the Schirmer test strip will be removed and the length of the tear absorption on the strip will be measured (millimeters/5 minutes)
Ocular Surface Disease Index (OSDI) score | Baseline, Day 14, Day 28, Day 56
  Change from Baseline in Ocular Surface Disease Index score. The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.
  The overall OSDI score defines the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.

SECONDARY OUTCOMES:
Tear Film Break-Up Time (TBUT) | Baseline, Day 14, Day 28, Day 56
  Change from Baseline in the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film. A TBUT greater than 15 seconds is considered normal, while a break time of less than 10 seconds is to be considered pathological.
Standard Patient Evaluation of Eye Dryness (SPEED) score | Baseline, Day 14, Day 28, Day 56
  Change from Baseline in the subjects' perception of eye dryness as assessed by Standard Patient Evaluation of Eye Dryness (SPEED) score.
  The SPEED questionnaire was designed in order to quickly track the progression of dry eye symptoms over time. This questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms. The symptoms assessed include dryness, grittiness, scratchiness, irritation, burning, watering, soreness, and eye fatigue. The questionnaire further assesses whether these symptoms were not problematic, tolerable, uncomfortable, bothersome, or intolerable
Corneal and Conjunctival Staining | Baseline, Day 56
  Change from Baseline in Corneal and Conjunctival Staining.
  Corneal and conjunctival staining of the ocular surface after instillation of vital dyes was developed to quantify epithelial surface damage in dry eye patients. A modified Oxford score is used to separately score cornea and conjunctiva from 0 to 5 (from 0 = none to 5 = extended areas of confluent stain).
Tear Osmolarity | Baseline, Day 56
  Change from Baseline in Tear Osmolarity
  Tear osmolarity refers to the amount of osmotically active particles. Tear osmolarity is abnormal at values greater than 300 milliosmole/L.
MMP-9 | Baseline, Day 56
  Change from Baseline in tear inflammatory marker MMP-9.
  InflammaDry MMP-9 test kits (QUIDEL, CA, USA) are used for qualitative determination of MMP-9 presence in both eyes. A positive MMP-9 result indicates the presence of MMP9 greater than or equal to 40 ng/ml, and a negative one indicates the presence of MMP-9 less than or equal to 40 ng/ml.
Rescue Medication Use | Baseline, Day 56
  Change from Baseline in rescue medication use

OTHER OUTCOMES:
Changes in White Blood Cell count | Baseline, Day 56
  Experimental outcome examining total White Blood Cell count via fasted whole blood samples
Changes in Red Blood Cell count | Baseline, Day 56
  Experimental outcome examining total Red Blood Cell count via fasted whole blood samples
Changes in Hemoglobin levels | Baseline, Day 56
  Experimental outcome examining total Hemoglobin via fasted whole blood samples
Changes in Hematocrit levels | Baseline, Day 56
  Experimental outcome examining total Hematocrit via fasted whole blood samples
Changes in Mean Corpuscular Volume | Baseline, Day 56
  Experimental outcome examining total Mean Corpuscular Volume via fasted whole blood samples
Changes in Mean Corpuscular Hemoglobin | Baseline, Day 56
  Experimental outcome examining total Mean Corpuscular Hemoglobin via fasted whole blood samples
Changes in Mean Corpuscular Hemoglobin Concentration | Baseline, Day 56
  Experimental outcome examining total Mean Corpuscular Hemoglobin Concentration via fasted whole blood samples
Changes in Red Cell Distribution Width | Baseline, Day 56
  Experimental outcome examining total Red Cell Distribution Width via fasted whole blood samples
Changes in Platelet Count | Baseline, Day 56
  Experimental outcome examining total Platelet count via fasted whole blood samples
Changes in Mean Platelet Volume | Baseline, Day 56
  Experimental outcome examining total Mean Platelet volume via fasted whole blood samples
Changes in Granulocyte levels | Baseline, Day 56
  Experimental outcome examining percentage of Granulocytes via fasted whole blood samples
Changes in Lymphocytes levels | Baseline, Day 56
  Experimental outcome examining percentage of Lymphocytes via fasted whole blood samples
Changes in Monocyte levels | Baseline, Day 56
  Experimental outcome examining percentage of Monocytes via fasted whole blood samples
Changes in Eosinophil levels | Baseline, Day 56
  Experimental outcome examining percentage of Eosinophil via fasted whole blood samples
Changes in Basophil levels | Baseline, Day 56
  Experimental outcome examining percentage of Basophil via fasted whole blood samples
Changes in Granulocyte count | Baseline, Day 56
  Experimental outcome examining total Granulocyte via fasted whole blood samples
Changes in Lymphocytes count | Baseline, Day 56
  Experimental outcome examining total Lymphocytes via fasted whole blood samples
Changes in Monocyte count | Baseline, Day 56
  Experimental outcome examining total Monocytes via fasted whole blood samples
Changes in Eosinophil count | Baseline, Day 56
  Experimental outcome examining total Eosinophil via fasted whole blood samples
Changes in Basophil count | Baseline, Day 56
  Experimental outcome examining total Basophil via fasted whole blood samples
Changes in Glucose levels | Baseline, Day 56
  Experimental outcome examining total Glucose via fasted whole blood samples
Changes in Blood Urea Nitrogen levels | Baseline, Day 56
  Experimental outcome examining total Blood Urea Nitrogen via fasted whole blood samples
Changes in Creatinine levels | Baseline, Day 56
  Experimental outcome examining total Serum Creatinine via fasted whole blood samples
Changes in Sodium levels | Baseline, Day 56
  Experimental outcome examining total Sodium via fasted whole blood samples
Changes in Potassium levels | Baseline, Day 56
  Experimental outcome examining total Potassium via fasted whole blood samples
Changes in Chloride levels | Baseline, Day 56
  Experimental outcome examining total Chloride via fasted whole blood samples
Changes in Carbon Dioxide levels | Baseline, Day 56
  Experimental outcome examining total Carbon Dioxide via fasted whole blood samples
Changes in Calcium levels | Baseline, Day 56
  Experimental outcome examining total Calcium via fasted whole blood samples
Changes in Total Protein levels | Baseline, Day 56
  Experimental outcome examining Total Protein via fasted whole blood samples
Changes in Albumin levels | Baseline, Day 56
  Experimental outcome examining total Albumin via fasted whole blood samples
Changes in Globulin levels | Baseline, Day 56
  Experimental outcome examining total Globulin via fasted whole blood samples
Changes in Total Bilirubin levels | Baseline, Day 56
  Experimental outcome examining total Bilirubin via fasted whole blood samples
Changes in Alkaline Phosphatase levels | Baseline, Day 56
  Experimental outcome examining total Alkaline Phosphatase via fasted whole blood samples
Changes in Alanine Transaminase levels | Baseline, Day 56
  Experimental outcome examining total Alanine Transaminase via fasted whole blood samples
Changes in Aspartate Aminotransferase levels | Baseline, Day 56
  Experimental outcome examining total Aspartate Aminotransferase via fasted whole blood samples
Changes in Albumin to Globulin ratio | Baseline, Day 56
  Experimental outcome examining the ratio of Albumin to Globulin via fasted whole blood samples
Changes in Blood Urea Nitrogen to Creatinine ratio | Baseline, Day 56
  Experimental outcome examining the ratio of Blood Urea Nitrogen to Creatinine via fasted whole blood samples
Changes in estimated Glomerular Filtration Rate | Baseline, Day 56
  Experimental outcome examining the Glomerular Filtration rate via fasted whole blood samples

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - True Eye Experts - Lutz, Lutz, Florida
  - Applied Science and Performance Institute, Tampa, Florida
  - True Eye Experts - New Tampa, Tampa, Florida

REFERENCES:
- [Derived] Gioia N, Gerson J, Ryan R, Barbour K, Poteet J, Jennings B, Sharp M, Lowery R, Wilson J, Morde A, Rai D, Padigaru M, Periman LM. A novel multi-ingredient supplement significantly improves ocular symptom severity and tear production in patients with dry eye disease: results from a randomized, placebo-controlled clinical trial. Front Ophthalmol (Lausanne). 2024 Apr 24;4:1362113. doi: 10.3389/fopht.2024.1362113. eCollection 2024. PMID 38984118